CLINICAL TRIAL: NCT01292369
Title: Observational Study Aimed to Characterize a System for Breast and Colon Cancer Diagnosis by Breath Testing - NaNose Study
Brief Title: Breath Testing for Breast and Colon Cancer Diagnosis- NaNose Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: NaNose LTD, AMIT- Alfred Mann institute in the technion
Other Study IDs: RMB-0566.CTIL
Record Dates: First submitted 2011-02-06; First posted 2011-02-09 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer; Colon Cancer
Keywords: breath test; colon cancer; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Breast cancer: Women diagnosed with breast cancer by a positive biopsy test after mammography.
- Breast control: Women with negative biopsy result done due to a suspicious mammography exam.
- Colon cancer: Men and women diagnosed with colon cancer by a positive colonoscopy and biopsy.
- Colon control: Men and women with negative colonoscopy and biopsy tested due to complaints indicating the possibility of colon cancer.

SUMMARY:
The concept of breath testing for various diseases has been around since ancient greece. It has been hypothesized that cancer is generating a unique pattern of compounds in patients' breath. This study is trying to characterize a novel system, based on nanoparticles technology, for cancer diagnosis through breath samples.

DETAILED DESCRIPTION:
Cancer is accompanied by increased oxidative stress and induction of polymorphic cytochrome P- 450 mixed oxidase enzymes (CYP). Both processes affect the abundance of volatile organic compounds (VOCs) in the breath because oxidative stress causes lipid peroxidation of polyunsaturated fatty acids in membranes, producing alkanes and methylalkanes which are catabolized by CYP.

In the Technion labs, a new system for breath samples diagnosis, is being developed. The system is based on Nanoparticles technology.

The current study will try to identify colon and breast cancer patients through their breath samples and discriminate them from healthy individuals.

Men and women coming for colonoscopy or breast biopsy will be recruited for the study. Breath samples will be taken from all volunteers before the medical test. Subjects with positive cancer results by biopsy will be the test groups for both diseases, all others will be the control.

The research goal is to test the NaNose system ability to discriminate between healthy and sick.

ELIGIBILITY:
Inclusion Criteria:

* Men and women attending Rambam medical center for either breast biopsy or colonoscopy.
* Suspicious finding on breast imaging requiring a biopsy.
* Complaints indicating the possibility of colon cancer: Blood in stool, weight loss, constipation, anemia, family history of colon cancer.

Exclusion Criteria:

* Other known active malignancy.
* History of malignant disease and treatments.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women coming for medical tests:
  1. Women coming for a breast biopsy following a suspicious breast imaging result.
  2. Men and women coming for a colonoscopy, reffered by their family physician, due to complaints indicating the possibility of colon cancer.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
System performance | 10 months
  Sensitivity and specificity of NaNose system in diagnosing cancer

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - RAMBAM medical center, Haifa
  - Carmel medical center, Haifa